CLINICAL TRIAL: NCT01940965
Title: An Open-Label, Multicenter 52-Week Study Assessing the Safety and Tolerability of Lixisenatide in Combination With Oral Anti-Diabetic Treatment in Patients With Type 2 Diabetes
Brief Title: Safety and Tolerability of Lixisenatide in Combination With Oral Anti-Diabetic Treatment in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS12809; U1111-1129-8754 (Other: UTN)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Biguanides; conotoxin GI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lixisenatide + Biguanide (Experimental): 52-week treatment with Lixisenatide in combination with biguanide (usual maintenance dose in the label)
  Interventions: Drug: lixisenatide AVE0010; Drug: biguanide
- Lixisenatide + TZD (Experimental): 52-week treatment with lixisenatide in combination with TZD (usual maintenance dose in the label)
  Interventions: Drug: lixisenatide AVE0010; Drug: TZD
- Lixisenatide + alpha-GI (Experimental): 52-week treatment with Lixisenatide in combination with alpha-GI (usual maintenance dose in the label)
  Interventions: Drug: lixisenatide AVE0010; Drug: alpha-GI
- Lixisenatide + Glinide (Experimental): 52-week treatment with Lixisenatide in combination with glinide (usual maintenance dose in the label)
  Interventions: Drug: lixisenatide AVE0010; Drug: glinide

INTERVENTIONS:
Drug: lixisenatide AVE0010 — Pharmaceutical form:solution Route of administration: Subcutaneous injection
Drug: biguanide — Pharmaceutical form:tablet Route of administration: oral
  Arms: Lixisenatide + Biguanide
Drug: TZD — Pharmaceutical form:tablet Route of administration: oral
  Arms: Lixisenatide + TZD
Drug: alpha-GI — Pharmaceutical form:tablet Route of administration: oral
  Arms: Lixisenatide + alpha-GI
Drug: glinide — Pharmaceutical form:tablet Route of administration: oral
  Arms: Lixisenatide + Glinide

SUMMARY:
Primary Objective:

The primary objective of this study is to assess the overall safety of lixisenatide once daily treatment in combination with background oral anti-diabetic treatment over 52 weeks in patients with type 2 diabetes in Japan.

Secondary Objective:

To assess the effects of lixisenatide in combination with background oral antidiabetic drug (OAD) on:

* HbA1c;
* Fasting plasma glucose;
* Body weight.

DETAILED DESCRIPTION:
54 weeks +/-11 days

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus diagnosed at least 1 year before the screening visit
* Patient treated for at least 3 months prior to screening visit with one of following OADs at a stable dose of at least usual maintenance dose as described in the label

  * a biguanide (metformin hydrochloride);
  * a thiazolidinedione (TZD) (pioglitazone hydrochloride);
  * an alpha-glucosidase inhibitor (alpha-GI) (acarbose, voglibose or miglitol);
  * or a glinide (nateglinide, repaglinide or mitiglinide);
* Signed written informed consent

Exclusion criteria:

* At screening HbA1c <7% or >9.5%;
* At screening: fasting plasma glucose >250 mg/dL (>13.9 mmol/L);
* Use of any glucose-lowering agent(s) other than the authorized patient's background treatment defined in I02 (as given in inclusion critieria) within 3 months prior to screening;
* Type 1 diabetes mellitus;
* Women of childbearing potential with no effective contraceptive method;
* Pregnancy or lactation;
* Laboratory findings at the time of screening:

  * Amylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN);
  * ALT >3 ULN;
* Any contra-indication to the patient's background oral anti-diabetic treatment;
* History of acute or chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease;
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes);
* Any previous treatment with lixisenatide (eg, participation in a previous study with lixisenatide) or any other GLP1 receptor agonist.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety over 52 weeks assessed by treatment emergent adverse event (TEAE), vital signs, 12-lead electrocardiogram (ECG), and laboratory data | 52 weeks

SECONDARY OUTCOMES:
Absolute change in HbA1c | From baseline to weeks 24 and 52
Absolute change in fasting plasma glucose | From baseline to weeks 24 and 52
Absolute change in body weight | From baseline to weeks 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- Japan (27):
  - Investigational Site Number 392335, Adachi-Ku
  - Investigational Site Number 392325, Chiba
  - Investigational Site Number 392328, Chiyoda-Ku
  - Investigational Site Number 392310, Chuoh-Ku
  - Investigational Site Number 392326, Chūōku
  - Investigational Site Number 392327, Chūōku
  - Investigational Site Number 392336, Kagoshima
  - Investigational Site Number 392314, Kamakura-Shi
  - Investigational Site Number 392334, Kashiwara-Shi
  - Investigational Site Number 392304, Kawagoe-Shi
  - Investigational Site Number 392306, Kawaguchi-Shi
  - Investigational Site Number 392307, Kisarazu-Shi
  - Investigational Site Number 392301, Koriyama-Shi
  - Investigational Site Number 392312, Mitaka-Shi
  - Investigational Site Number 392302, Mito
  - Investigational Site Number 392324, Mito
  - Investigational Site Number 392331, Nagoya
  - Investigational Site Number 392332, Nagoya
  - Investigational Site Number 392329, Ohta-Ku
  - Investigational Site Number 392322, Okawa-Shi
  - Investigational Site Number 392333, Osaka
  - Investigational Site Number 392330, Sagamihara-Shi
  - Investigational Site Number 392320, Saijo-Shi
  - Investigational Site Number 392303, Sakado-Shi
  - Investigational Site Number 392311, Shinjuku-Ku
  - Investigational Site Number 392316, Shizuoka
  - Investigational Site Number 392319, Suita-Shi